CLINICAL TRIAL: NCT00123643
Title: Comparison of Rosiglitazone Versus Glyburide on Vascular Structure and Function in Type 2 Diabetic Patients
Brief Title: Vascular Effects of Rosiglitazone Versus Glyburide in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Paul Heart Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Aaron S. Kelly, Ph.D., Assistant Professor, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GSK2002-2
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: thiazolidinedione; sulfonylurea; endothelial function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone (Experimental)
  Interventions: Drug: rosiglitazone
- Glyburide (Active Comparator)
  Interventions: Drug: glyburide

INTERVENTIONS:
Drug: rosiglitazone
  Arms: Rosiglitazone
Drug: glyburide
  Arms: Glyburide

SUMMARY:
The purpose of this study is to compare the vascular effects of two commonly used diabetes medications, rosiglitazone and glyburide in type 2 diabetic patients.

DETAILED DESCRIPTION:
Rosiglitazone and glyburide are two commonly used diabetic medications that have both been shown to be effective in controlling blood glucose levels. Since they work in different ways, they may have different effects on the health of the blood vessels. This study will assess which medication is better at improving the health of the arteries separate from the blood glucose lowering effects. Artery health will be assessed non-invasively by ultrasound. Certain markers of atherosclerosis found in the blood will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-75 years
* Type 2 diabetes mellitus for less than or equal to 10 years
* Pre-screening HbA1c > 6.5 %
* Screening 110 mg/dl < fasting plasma glucose < 240 mg/dl after 2 weeks of metformin 500 mg twice daily (b.i.d.)

Exclusion Criteria:

* Thiazolidinedione or sulfonylurea use in previous 30 days (may undergo washout period of 30 days)
* Known contraindications to use of thiazolidinedione or sulfonylurea
* Female patients must be postmenopausal, surgically sterile, or using adequate contraception
* Uncontrolled hyperlipidemia according to American Heart Association (AHA) guidelines
* Subcutaneous insulin use
* Elevated liver enzymes (2.5 times the upper limit of the reference range)
* Serum creatinine >160 mmol/l
* Anemia (Hb <11 g/dl for men or <10 g/dl for women)
* Body mass index (BMI) <22 or >42 kg/m2
* History of ketoacidosis
* Angina/New York Health Academy class III/IV cardiac insufficiency
* Electrocardiographic evidence of marked left ventricular hypertrophy
* Uncontrolled hypertension according to AHA guidelines
* Hemoglobinopathy

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Bank, M.D., Principal Investigator — St. Paul Heart Clinic
Locations (1):
- St. Paul Heart Clinic, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment was performed at medical clinics
Pre-assignment Details: patients taking thiazolidinediones or sulfonylureas were allowed to washout of these medications 30 days prior to randomization
Period: Overall Study
Arm/Group | Rosiglitazone | Glyburide
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Glyburide | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 8 | 24
  >=65 years | 4 | 8 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 57.9 (8.2) | 63.1 (7.8) | 60.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation
Description: Measure of endothelial function
Time Frame: change from baseline to 6 months
Population: All completers were analyzed
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rosiglitazone | Glyburide
Number analyzed (Participants) | 20 | 16
percent change | 6.8 (3.7) | 5.5 (3.1)

ADVERSE EVENTS:
Time Frame: 6-months
Arm/Group | Rosiglitazone | Glyburide
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/16

LIMITATIONS AND CAVEATS:
Small sample size; unbalanced sex distribution between groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No